CLINICAL TRIAL: NCT05747859
Title: Voice Telerehabilitation for Patients Affected by Iatrogenic Unilateral Vocal Fold Paralysis: From Necessity to Opportunity in the COVID-19 Time
Brief Title: Voice Telerehabilitation
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, mari Giorgia, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4427
Record Dates: First submitted 2023-02-15; First posted 2023-02-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Vocal Fold Palsy
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: teletherapy — speech therapy remotely delivered

SUMMARY:
The aim of the study was to determine functional results of telerehabilitation (TR) in subjects affected by iatrogenic unilateral vocal fold paralysis (UVFP) during the COVID-19 pandemic outbreak. 40 patients with iatrogenic unilateral vocal fold paralysis underwent voice teletherapy with a synchronous approach. A multidimensional assessment by means of videolaryngostroboscopy, acoustic and perceptual analysis and patient self-assessment was carried out before, at the end of teletherapy and six months later.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-75 years
* onset of UVFP less than 1 month before
* internet access
* availability and ability to use a computer with an internal or external webcam.

Exclusion Criteria:

* previous history of laryngeal pulmonary or gastric surgery
* current or previous pulmonary diseases
* hearing loss, neurological or motor deficits
* reading difficulties
* dysphagia
* unavailability of a computer and a webcam.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 subjects affected by permanent iatrogenic UVFP
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
analysis | 1 month
  to analyze the functional outcomes achieved by a group of patients with recent onset of iatrogenic UVFP who were referred to TR using a synchronous approach.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgia Mari, SLP MSC, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No